CLINICAL TRIAL: NCT04985695
Title: Influence of Analgesic Technique on Post Operative Rehabilitation After Median Laparotomy: Comparison Between Thoracic Epidural Anesthesia Versus Bilateral Rectus Sheath Block
Brief Title: Influence of Analgesic Technique on Post Operative Rehabilitation After Median Laparotomy
Acronym: QORRECTCATH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-01-CHRMT
Record Dates: First submitted 2021-07-08; First posted 2021-08-02 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-10

CONDITIONS: Laparotomy
Keywords: postoperative rehabilitation
MeSH Terms: interventions — Analgesia, Epidural; Laparotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic epidural anesthesia (Active Comparator): Epidural analgesia during midline laparotomy
  Interventions: Drug: Epidural analgesia; Procedure: Laparotomy
- Bilateral rectus sheath block (Experimental): Bilateral rectus sheath block during midline laparotomy
  Interventions: Drug: Bilateral rectus sheath block; Procedure: Laparotomy

INTERVENTIONS:
Drug: Epidural analgesia — All patients received local anesthesia (3-5 ml of 2% Lidocaine). During the preoperative induction of anaesthesia a catheter was inserted 4cm into the epidural space. The catheter will be load during the intervention (0.1 ml/kg/h). In postoperative situation, a patient controlled epidural analgesia was introduced with a debit adapted to the arterial pressure.
  Arms: Thoracic epidural anesthesia
Drug: Bilateral rectus sheath block — Bilateral rectus sheath block was performed Under general anesthesia and with ultrasound guidance. Rectus sheath block was inserted on each side of the abdomen. All patients received ropivacaine through elastomeric pump
  Arms: Bilateral rectus sheath block
Procedure: Laparotomy — A midline sub or supra umbilical laparotomy or xypho-pubian laparotomy

SUMMARY:
Randomized controlled trial (1:1) in two parallel groups, multicentric, open-label, comparing two locoregional anesthesia (LRA) techniques as integral parts of multimodal analgesia: the control group will benefit from epidural anesthesia, while the experimental group will benefit from bilateral placement of catheters in the sheath of the rectus abdominis muscles.

DETAILED DESCRIPTION:
Implementation of fast-track rehabilitation surgery was essential in patient care, specially in oncological point.

In this way, uses of the technic of local anesthesia, include epidural analgesia, was essential, but this one is associated with few complications. Emergence of new technic of anesthesia with a comparative analgesia and without side effects should be a better alternative than epidural analgesia. Thus, bilateral rectus sheath block has been reported to be effective in management of postoperative pain.

After signing of the informed consent, two postoperative analgesia techniques were investigated in patients undergoing midline laparotomy.

The main objective of this study is to compare the influence of analgesic technique on the Quality of Recovery-15 score. The study design was a prospective, randomized trial with 2 parallel arms (epidural analgesia vs bilateral rectus sheath block).

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) Class I-IV adult, with programmed midline laparotomy
* Have given an informed written consent
* Able to read and understand french language
* Affiliation to a social security system

Exclusion Criteria:

* Local anesthesic contraindication (allergy, porphyria, haemolytic anaemia, uncontrolled epilepsy, or severe cardiac conduction disorders) or TEA (coagulation disorders, progressive neurological disease, or severe spinal disorder),
* Epidural analgesia contraindication
* With impossibility to set up bilateral rectus sheath block
* Participation in another clinical study
* Pregnant women
* Patients deprived of their liberty by a judicial or administrative decision,
* Patients undergoing psychiatric care under articles L.3212-1 and L.3213-1 of the French Public Health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2028-10-10 (Estimated); Study Completion 2029-04-10 (Estimated)

PRIMARY OUTCOMES:
Change in total QoR-15 score | Postoperative day 2
  The Quality of Recovery-15 (QoR-15) included five dimensions: physical comfort, emotional state, pain, psychological support and physical independence. Each item was assessed using an 11-point numerical rating scale (for positive itel, 0="none of the time" to 10="all the time"; for negative items the scoring was reversed).

SECONDARY OUTCOMES:
Change in total Qor-15 score on postoperative days 1 and 3 compared to the day before surgery | Postoperative days 1, and 3
  The Quality of Recovery-15 (QoR-15) included five dimensions: physical comfort, emotional state, pain, psychological support and physical independence. Each item was assessed using an 11-point numerical rating scale (for positive itel, 0="none of the time" to 10="all the time"; for negative items the scoring was reversed).
Efficacy of postoperative analgesia | Day 0 and Postoperative days 1, 2, 3 and 30
  The efficacy of postoperative analgesia was compared between the two groups with the visual analog scale (VAS). The VAS intensity rating consisted of a 100-mm line with the end points no pain (0 mm) and worst pain (100 mm). Study participants were asked to evaluated with a mark on the line their current pain intensity. The difference between each postoperative treatment VAS score was compared.
Impact of arterial hypotension | Postoperative days 1, 2 and 3
  The impact of arterial hypotension was compared between the two groups with the arterial pressure value before and after laparotomy
Impact of orthostatic hypotension | Postoperative days 1, 2 and 3
  The impact of orthostatic hypotension was compared between the two groups with the arterial pressure value before and after surgery.
Occurrence of nausea and/or vomiting | Day 0, Postoperative days 1, 2 and 3 and at hospital discharge up to 30 days
  The effect of analgesic technique on nausea and/or vomiting is calculated on the basis of the number of anti-vomiting prescribed.
Postoperative complications link to analgesic technique | Postoperative days 1, 2 and 3
  Number of postoperative complication in both groups
The length of stay | at hospital discharge up to 30 days
  Comparison of the length of stay between the two groups
Return to normal bowel function | Postoperative days 1, 2 and 3 and at hospital discharge up to 30 days
  Delay in hours to promotes normal digestive activity. The included the times to recovery the first bowel sounds, first anal exhaust and defecation.
The quantity of morphine or equivalent | Day 0 and Postoperative days 1, 2 and 3
  The quantity of morphine or equivalent administered during the 48 first hours in both groups
Urinary catheterization | at hospital discharge up to 30 days
  The time during which the patients are taking recourse to postoperative urinary catheterization
Total distance covered | Postoperative days 1, 2 and 3
  Compare the impact of postoperative analgesia in Walking distance (meter) within days following the operation
Failure to set up a catheter | Postoperative day 1
  Number of Failure to delivery catheter in both techniques
The time until the first raised | Postoperative days 1, 2 and 3 and at hospital discharge up to 30 days
  Delay before the first raised in hours
Impact of premature discontinuation of local anesthetic perfusion | on day 0
  Number of premature discontinuation of local anesthetics
Patient satisfaction and need for further consultation | at hospital discharge up to 30 days and on postoperative day 30
  Satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BECRET, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (2):
- France (2):
  - CHR Metz Thionville Hopital de Mercy, Metz, Moselle
  - CHR Metz-Thionville Hopital Bel Air, Thionville

IPD SHARING:
Plan to Share IPD: No
According to the French law and the French Data Protection Authority (CNIL), we won't be able to publicly share individual participant data, but we plan to share their conclusions through peer-reviewed publications and conferences.

REFERENCES:
- [Derived] Maury T, Elnar A, Marchionni S, Frisoni R, Goetz C, Becret A. Effect of rectus sheath anaesthesia versus thoracic epidural analgesia on postoperative recovery quality after elective open abdominal surgery in a French regional hospital: the study protocol of a randomised controlled QoR-RECT-CATH trial. BMJ Open. 2023 May 23;13(5):e069736. doi: 10.1136/bmjopen-2022-069736. PMID 37221022